CLINICAL TRIAL: NCT03501589
Title: Molecular Modulation of the Growth Plate
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, A. Noelle Larson, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 13-005403
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Growth Plate Injury
MeSH Terms: conditions — Salter-Harris Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Growth plate cartilage or bone removed as a normal part of surgical procedure that would otherwise be disposed of as waste tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The researchers are trying to identify molecular mechanisms that control growth plate mediated limb growth and identify agents that can be used to enhance or slow growth.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally immature children/adults undergoing surgical procedures where growth plate cartilage is removed as a normal part of their procedure; or patients undergoing surgical procedures where bone is removed as a normal part of their procedure.

Exclusion Criteria:

* Skeletally mature children/adults

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery where growth plate cartilage or bone is removed as discarded tissue, waste, or surgical debris.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
RNA expression | End of Study (1/2019
  Measure RNA levels in growth plate tissue samples (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: A. Noelle Larson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic', Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials